CLINICAL TRIAL: NCT00927563
Title: Tolcapone Treatment of Pathological Gambling: An Open-Label Study
Brief Title: Tolcapone Treatment of Pathological Gambling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901M58441
Record Dates: First submitted 2009-06-12; First posted 2009-06-25 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Pathological Gambling
Keywords: Gambling; Addiction
MeSH Terms: conditions — Gambling; Behavior, Addictive | interventions — Tolcapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tolcapone (Experimental): Tolcapone 100-300mg/day
  Interventions: Drug: Tolcapone

INTERVENTIONS:
Drug: Tolcapone — pill, 100-300mg/day for 8 weeks
  Other Names: Brand name: TASMAR

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of tolcapone in pathological gambling.

DETAILED DESCRIPTION:
The proposed study will consist of 8 weeks of treatment with tolcapone in 10 subjects with pathological gambling. The hypothesis to be tested is that tolcapone will be effective in reducing the urges to gamble in patients with pathological gambling. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 21-75;
2. Meet diagnostic criteria for current pathological gambling based on DSM-IV criteria and confirmed using the clinician-administered Structured Clinical Interview for Pathological Gambling (SCI-PG) (Grant et al., 2004);
3. Gambling behavior within 2 weeks prior to enrollment;
4. Women of child bearing age are required to have a negative result on a beta-human chorionic gonadotropin pregnancy test;
5. Women of childbearing potential utilizing a medically accepted form of contraception defined as double barrier, oral contraceptive, injectable contraceptive, implantable contraceptive devices, and abstinence.

Exclusion Criteria:

1. Infrequent gambling (i.e. less than one time per week) that does not meet DSM-IV criteria for PG;
2. Unstable medical illness or clinically significant abnormalities on laboratory tests, EKG, or physical examination at screen as determined by the investigator;
3. History of elevated liver enzymes (AST/ALT) or other liver abnormalities;
4. History of seizures;
5. Myocardial infarction within 6 months;
6. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
7. A need for medication other than tolcapone with possible psychotropic effects or unfavorable interactions as determined by the investigator;
8. Clinically significant suicidality (defined as score 2 or higher on HAM-D item 3);
9. Current co-morbid Axis I disorder determined by the Structured Clinical Interview for DSM-IV (SCID), (First et al., 1995) - except for nicotine dependence;
10. Lifetime history of bipolar disorder type I or II, schizophrenia, or any psychotic disorder determined by SCID;
11. Clinically significant cognitive impairment (defined as score less than 88 on 3MS);
12. Current or recent (past 3 months) DSM-IV substance abuse or dependence;
13. Positive urine drug screen at screening;
14. Initiation of psychotherapy or behavior therapy for pathological gambling within 3 months prior to study baseline;
15. Previous treatment with tolcapone;
16. Treatment with an investigational medication or depot neuroleptics within 3 months;
17. Refusal to sign the tolcapone information sheet.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, Principal Investigator — University of Minnesota
Locations (1):
- Ambulatory Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Grant JE, Odlaug BL, Chamberlain SR, Hampshire A, Schreiber LR, Kim SW. A proof of concept study of tolcapone for pathological gambling: relationships with COMT genotype and brain activation. Eur Neuropsychopharmacol. 2013 Nov;23(11):1587-96. doi: 10.1016/j.euroneuro.2013.07.008. Epub 2013 Aug 6. PMID 23953269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via media advertisement from January 2010 through February 2012 at the University of Minnesota Department of Psychiatry.
Pre-assignment Details: Subjects could not be using concomitant use of psychotropic medications with possible effects on PG symptoms (i.e. antidepressants, opioid antagonists)(due to possible interference of results) or have had previous treatment with tolcapone.
Groups:
- Tolcapone: Tolcapone 100-300mg/day
  Tolcapone : pill, 100-300mg/day for 8 weeks
Period: Overall Study
Arm/Group | Tolcapone
Started | 24
Completed | 22
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tolcapone
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Scale (CGI)
Description: The overall impression of the clinician of the severity of the subject. Scores between 1 and 7 with 1 not being ill at all and 7 being one of the worst cases seen. CGI is assessed at every visit (1-5), but only the final visit will be reported here.
Time Frame: Visit 5 (final visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolcapone
Number analyzed (Participants) | 22
units on a scale | 2.88 (1.30)

2. Secondary Outcome: Yale Brown Obsessive Compulsive Scale Modified for Pathological Gambling (PG-YBOCS)
Description: Scale used to measure severity of gambling. Scores could range from 0-40 with 0 being the least severe and 40 being the most severe. Here the total score was used. The PG-YBOCS was completed at every visit (1-5), but the final visit (visit 5) will be the only score reported.
Time Frame: Visit 5 (final visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolcapone
Number analyzed (Participants) | 22
units on a scale | 10.50 (7.02)

3. Secondary Outcome: Gambling Symptom Assessment Scale (G-SAS)
Description: Self report test of severity of gambling on a scale from 0-48 with 48 being the most severe. The G-SAS was performed at every visit (1-5), but only the final visit (visit 5) will be reported here as a final score.
Time Frame: Visit 5 (final visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolcapone
Number analyzed (Participants) | 22
units on a scale | 18.67 (10.58)

ADVERSE EVENTS:
Arm/Group | Tolcapone
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolcapone (N=24)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dry Mouth (Skin and subcutaneous tissue disorders) | 2 (2)
Vivid Dreams (Psychiatric disorders) | 2 (2)
Broken Sleep (Psychiatric disorders) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 1 (1)
Headache (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study did not assess treatment effects beyond an 8-week treatment period and these results may not generalize to the larger population of people with PG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No